CLINICAL TRIAL: NCT02540109
Title: Targeted Transcranial Electrotherapy for Stroke Rehabilitation - Exploratory Trial on Aphasia
Brief Title: Targeted Electrotherapy for Aphasia Stroke Rehabilitation (TEASER) - Phase II Multi-Center Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soterix Medical (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Georgetown University (Other); University of North Carolina, Chapel Hill (Other); The City College of New York (Other); Medstar Health Research Institute (Other); University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMI092144-P2; 1R44NS092144 (NIH)
Record Dates: First submitted 2015-08-31; First posted 2015-09-03 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Chronic Aphasia
Keywords: Stroke; Anomia
MeSH Terms: conditions — Stroke; Anomia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-Definition tDCS (Active) (Experimental)
  Interventions: Device: HD-tDCS (Soterix Medical, Active)
- High-Definition tDCS (Sham) (Experimental)
  Interventions: Device: HD-tDCS (Soterix Medical, Sham)

INTERVENTIONS:
Device: HD-tDCS (Soterix Medical, Active) — Subject will be given individualized dose (number of electrodes and electrode placement) through High-Definition electrodes to target fMRI determined targets.
  Other Names: Soterix Medical High-Definition MxN stimulator; Soterix Medical HDTargets
  Arms: High-Definition tDCS (Active)
Device: HD-tDCS (Soterix Medical, Sham) — Subject will be given individualized dose (number of electrodes and electrode placement) through High-Definition electrodes to target fMRI determined targets.
  Other Names: Soterix Medical High-Definition MxN stimulator; Soterix Medical HDTargets
  Arms: High-Definition tDCS (Sham)

SUMMARY:
This Phase II study aims to ascertain the effectiveness of HD-tDCS for adjunctive treatment of anomia in chronic aphasia post stroke. Furthermore, it will help explore factors such as alternate outcome measures, subject selection criteria, and benefits of extended treatment duration. These results will be compared to an existing trial using conventional non-targeted tDCS with the same design and outcomes. Patients will be treated with HD-tDCS while performing computerized anomia treatment. The basis behind this method is that language therapy is mediated by cortical areas that are most effectively activated during the training tasks, thus increasing electric stimulation in these areas may improve learning outcomes. To better understand the long term benefits of the adjunctive treatment, patients will be screened again four weeks and six months after study using the same anomia tests. If HD-tDCS shows promising results in increasing the learning outcomes of anomia treatment, a Phase III trial can be considered.

ELIGIBILITY:
Inclusion Criteria:

* one-time ischemic stroke in the left hemisphere
* greater than 6-months post-stroke onset
* between 25 and 75 years of age
* aphasia diagnosis (as determined by pre-treatment language-based testing)
* right-handed (before the stroke)
* native speaker of English
* ability to provide informed written or verbal consent

Exclusion Criteria:

* clinically reported history of dementia, alcohol abuse, psychiatric disorder, traumatic brain injury, or extensive visual acuity or visual-spatial problems
* factors contraindicative of tDCS administration (sensitive scalp, previous brain surgery)
* prior history of epileptic or unprovoked seizures occurring during the previous 12 months.
* Presence of Metal implants of claustrophobia (not able to undergo MRI)
* Pregnancy
* Presence of any other neurological disease than stroke
* Childhood history of speech, language, hearing, or intellectual impairment

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Effect size of HD-tDCS for the adjunctive treatment of anomia in chronic aphasia after stroke | 3 weeks
  The primary outcome measures the ability of subjects to name objects in a standardized naming task. Prior to treatment MRI and fMRI are acquired to inform the individualized current flow models for optimal targeting.

SECONDARY OUTCOMES:
Determine alternate outcome measures | 4 weeks and 6 months follow up
  Determine alternate outcome measures, such as naming performance at 4 weeks and 6 months after treatment and improvements in more general discourse performance. An additional secondary exploratory objective is to perform a screening comparison of HD-tDCS with historical data on conventional non-targeted tDCS using sponge electrodes.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Datta, Ph.D, Study Chair — Soterix Medical Inc.; Lucas C Parra, Ph.D, Study Chair — City University of New York - CCNY
Locations (2):
- United States (2):
  - Georgetown University Medical Center (Peter Turkeltaub, MD, Ph.D.), Washington D.C., District of Columbia
  - University of North Carolina School of Medicine (Adam Jacks, Ph.D.), Chapel Hill, North Carolina

REFERENCES:
- See also: Feasibility of using high-definition transcranial direct current stimulation (HD-tDCS) to enhance treatment outcomes in persons with aphasia. — http://www.ncbi.nlm.nih.gov/pubmed/25547776